CLINICAL TRIAL: NCT06528340
Title: Study of Pregnancies Outcomes in Advanced Maternal Age Women
Brief Title: Pregnancies Outcomes in Advanced Maternal Age Women
Acronym: POIAMA
Status: Completed | Type: Observational
Sponsor: Centro di Ricerca Clinica Salentino (Network)
Responsible Party: Sponsor
Other Study IDs: CER 0424
Record Dates: First submitted 2024-06-21; First posted 2024-07-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Maternal Age Pregnancy; Premature; Labor Complication; Delivery Complication; Delivery Complications Affecting Fetus / Newborn; Delivery;Complicated;Liveborn; Cesarean Section Complications; Complication of Labor and Delivery
Keywords: Advanced maternal age; Pregnancy outcomes; Delivery; Labor; Uterine ageing; Cesarean section complications; Operative delivery complications; Female reproductive ageing
MeSH Terms: conditions — Premature Birth; Obstetric Labor Complications | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: spontaneous delivery — The women will be followed until the birth, in which the 3 traditional 3 methods will be carried out (spontaneous, vaginal operating, abdominal operation)
  Other Names: operative delivery; cesarean section

SUMMARY:
Pregnancies occurring in advanced maternal age (AMA) have become more common over the last few decades for a variety of reasons. Prominent contributor to this trend are the significant advancement in assisted reproductive technology (ART) and the growing accessibility to egg donation. Delaying having children is generally associated with other variables, such as the availability of various forms of contraception, which have decreased the number of unintended births and given women more autonomy over when they choose to become pregnant. In addition, from a socioeconomic standpoint, greater education and career options for women are major contributors to this phenomenon. Women with postsecondary education are especially affected by this issue since they are more likely to miss out on professional opportunities, money, and social standing when they become mothers. Studies show that women with a tertiary level of education stay pregnant later in life, compared to women with a lower level of education. Moreover, severe economic volatility throughout the early adult years, delays in the establishment of partnerships and marriages, and the shift from family homes to independent living all serve to worsen the tendency. In this investigation, we will seek, with a critical eye, to evaluate the implications of a pregnant woman in AMA and her outcomes, trying to highlight all the possible complications and problems of a pregnancy in AMA, with an evaluation of a big volume of AMA women in pregnancy and at delivery.

DETAILED DESCRIPTION:
Aims:

1. Primary aim is to investigate outcomes of pregnancies in advanced maternal age, in relation to maternal morbidity
2. Secondary aim is to investigate neonatal outcomes of pregnancies in advanced maternal age
3. Third aim is to evaluate if the pregnancy outcomes differ in relation to conception (spontaneous, IVF/ET, IVF/DO/ET or CRYO) INCLUSION CRITERIA

1. pregnants older than 45 yrs at the time of delivery, regardless mode of conception 2. gestational age ≥24 weeks of gestation EXCLUSION CRITERIA

1. missing data relevant for the study
2. surrogacy MATERIALS AND METHODS The study will be conducted as multicentric observational study including both vaginal and cesarean section deliveries in each participating center from January 1st 2019 until December 31st, 2025 (period of seven years). In each participating center, one person will be in charge for data collection and filling the SPSS database after obtaining the approval of the local Ethic Committee. As the study is observational and all the procedures will be conducted according to the local practice, informed consent from patients is not necessary.

Following data collection and termination of the study, a single researcher will oversee the SPSS data collection for all the participating centers, checking the quality of data and submitting it for statistical analysis.

The following data will be collected for each patient:

1. maternal age at delivery
2. gravidity
3. parity
4. gestational age at delivery
5. data about conception: spontaneous, IVF, oocyte donation
6. use of cryopreserved material
7. maternal comorbidity
8. maternal pregnancy complication
9. use of prenatal diagnostics
10. mode od delivery
11. neonatal weight and AS
12. presence of fetal anomalies
13. IUGR
14. placental pathology: previa, abruption, abnormally invasive placenta
15. peripartum hemorrhage
16. ICU treatment after delivery
17. duration of postpartum hospital treatment in days
18. prolonged postpartum hospitalization peripartum major complications (hysterectomy, hematoma, relaparotomy, ligation of major blood vessels (uterine, ovarian, iliac), etc.)

ELIGIBILITY:
Inclusion Criteria:

1. pregnants older than 45 yrs at the time of delivery, regardless mode of conception
2. gestational age ≥24 weeks of gestation

Exclusion Criteria:

1. missing data relevant for the study
2. surrogacy

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women in Advanced Maternal Age will be enrolled for the study, in order to better understand the outcomes of pregnancy. They are all healthy women, in spontaneous pregnancy or assisted by fertilization techniques.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcomes | 1 year
  To investigate outcomes of pregnancies in advanced maternal age, in relation to maternal morbidity, as complications in pregnancy, gestational age at delivery, type of delivery, maternal pregnancy complications, placental pathology, peripartum hemorrages, duration of hospital stay, prolonged hospitalization, peripartum major complications, etc

SECONDARY OUTCOMES:
Perinatal outcomes | 1 year
  The results of this study will show whether maternal age has a significant association with preterm birth.
Perinatal outcomes | 1 year
  The results of this study will show whether maternal age has a significant association with low birth weight
Perinatal outcomes | 1 year
  The results of this study will show whether maternal age has a significant association with low fifth-minute Apgar score
Perinatal outcomes | 1 year
  The results of this study will show whether maternal age has a significant association with perinatal death.

OTHER OUTCOMES:
Outcomes based on type of conception | 1 year
  To evaluate if the pregnancy outcomes in AMA women differ in relation to conception (if spontaneous, or by IVF/ET, by IVF/DO/ET or by CRYO).

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA TINELLI, MD, Study Chair — Ospedale Veris delli Ponti, Scorrano, Le
Locations (1):
- Ospedale Veris delli Ponti, Scorrano, Lecce, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Friese C, Becker G, Nachtigall RD. Older Motherhood and the Changing Life Course in the Era of Assisted Reproductive Technologies. J Aging Stud. 2008 Jan;22(1):65-73. doi: 10.1016/j.jaging.2007.05.009. PMID 18443646
- [Result] Ubaldi FM, Cimadomo D, Vaiarelli A, Fabozzi G, Venturella R, Maggiulli R, Mazzilli R, Ferrero S, Palagiano A, Rienzi L. Advanced Maternal Age in IVF: Still a Challenge? The Present and the Future of Its Treatment. Front Endocrinol (Lausanne). 2019 Feb 20;10:94. doi: 10.3389/fendo.2019.00094. eCollection 2019. PMID 30842755
- [Result] Glick I, Kadish E, Rottenstreich M. Management of Pregnancy in Women of Advanced Maternal Age: Improving Outcomes for Mother and Baby. Int J Womens Health. 2021 Aug 10;13:751-759. doi: 10.2147/IJWH.S283216. eCollection 2021. PMID 34408501
- [Result] Traisrisilp K, Tongsong T. Pregnancy outcomes of mothers with very advanced maternal age (40 years or more). J Med Assoc Thai. 2015 Feb;98(2):117-22. PMID 25842790
- [Result] Mathews TJ, Hamilton BE. Mean Age of Mothers is on the Rise: United States, 2000-2014. NCHS Data Brief. 2016 Jan;(232):1-8. PMID 26828319
- [Result] Zhu C, Zhang S, Shen L, Ye L, Zhan M, Cai S, Huang J, Wang Z, Chen H. Changes in the characteristics and outcomes of high-risk pregnant women who delivered prior to and after China's universal two-child policy: a real-world retrospective study, 2010-2021. BMC Public Health. 2024 Jan 31;24(1):336. doi: 10.1186/s12889-024-17810-9. PMID 38297279
- [Result] Goisis A. How Are Children of Older Mothers Doing? Evidence from the United Kingdom. Biodemography Soc Biol. 2015;61(3):231-51. doi: 10.1080/19485565.2014.1001887. PMID 26652679
- [Result] Myrskyla M, Barclay K, Goisis A. Advantages of later motherhood. Gynakologe. 2017;50(10):767-772. doi: 10.1007/s00129-017-4124-1. Epub 2017 Aug 29. PMID 29070913
- [Result] Broekmans FJ, Knauff EA, te Velde ER, Macklon NS, Fauser BC. Female reproductive ageing: current knowledge and future trends. Trends Endocrinol Metab. 2007 Mar;18(2):58-65. doi: 10.1016/j.tem.2007.01.004. Epub 2007 Feb 1. PMID 17275321
- [Result] Charalambous C, Webster A, Schuh M. Aneuploidy in mammalian oocytes and the impact of maternal ageing. Nat Rev Mol Cell Biol. 2023 Jan;24(1):27-44. doi: 10.1038/s41580-022-00517-3. Epub 2022 Sep 6. PMID 36068367
- [Result] Baird DT, Collins J, Egozcue J, Evers LH, Gianaroli L, Leridon H, Sunde A, Templeton A, Van Steirteghem A, Cohen J, Crosignani PG, Devroey P, Diedrich K, Fauser BC, Fraser L, Glasier A, Liebaers I, Mautone G, Penney G, Tarlatzis B; ESHRE Capri Workshop Group. Fertility and ageing. Hum Reprod Update. 2005 May-Jun;11(3):261-76. doi: 10.1093/humupd/dmi006. Epub 2005 Apr 14. PMID 15831503
- [Result] Hall JE. Neuroendocrine changes with reproductive aging in women. Semin Reprod Med. 2007 Sep;25(5):344-51. doi: 10.1055/s-2007-984740. PMID 17710730
- [Result] Tinelli A, Andjic M, Morciano A, Pecorella G, Malvasi A, D'Amato A, Sparic R. Uterine Aging and Reproduction: Dealing with a Puzzle Biologic Topic. Int J Mol Sci. 2023 Dec 25;25(1):322. doi: 10.3390/ijms25010322. PMID 38203493
- [Result] Kosmas IP, Malvasi A, Vergara D, Mynbaev OA, Sparic R, Tinelli A. Adrenergic and Cholinergic Uterine Innervation and the Impact on Reproduction in Aged Women. Curr Pharm Des. 2020;26(3):358-362. doi: 10.2174/1381612826666200128092256. PMID 32003664
- [Result] Tinelli A. Editorial (Thematic Issue: Uterine Innervation and Clinical Features in Obstetrics & Gynecology). Curr Protein Pept Sci. 2017;18(2):106-107. doi: 10.2174/138920371802161215213813. No abstract available. PMID 28430090
- [Result] Tinelli A, Malvasi A, Rahimi S, Negro R, Vergara D, Martignago R, Pellegrino M, Cavallotti C. Age-related pelvic floor modifications and prolapse risk factors in postmenopausal women. Menopause. 2010 Jan-Feb;17(1):204-12. doi: 10.1097/gme.0b013e3181b0c2ae. PMID 19629013
- [Result] Tinelli A, Vergara D, Ma Y, Malvasi A. Dystocia, Uterine Healing and Uterine Innervation: An Unexplored Intersection. Curr Protein Pept Sci. 2020;21(5):440-442. doi: 10.2174/1389203720666190717115744. No abstract available. PMID 32268856
- [Result] Frick AP. Advanced maternal age and adverse pregnancy outcomes. Best Pract Res Clin Obstet Gynaecol. 2021 Jan;70:92-100. doi: 10.1016/j.bpobgyn.2020.07.005. Epub 2020 Jul 15. PMID 32741623
- [Result] Radon-Pokracka M, Adrianowicz B, Plonka M, Danil P, Nowak M, Huras H. Evaluation of Pregnancy Outcomes at Advanced Maternal Age. Open Access Maced J Med Sci. 2019 Jun 30;7(12):1951-1956. doi: 10.3889/oamjms.2019.587. eCollection 2019 Jun 30. PMID 31406535
- [Result] Kahveci B, Melekoglu R, Evruke IC, Cetin C. The effect of advanced maternal age on perinatal outcomes in nulliparous singleton pregnancies. BMC Pregnancy Childbirth. 2018 Aug 22;18(1):343. doi: 10.1186/s12884-018-1984-x. PMID 30134873
- [Result] Kenny LC, Lavender T, McNamee R, O'Neill SM, Mills T, Khashan AS. Advanced maternal age and adverse pregnancy outcome: evidence from a large contemporary cohort. PLoS One. 2013;8(2):e56583. doi: 10.1371/journal.pone.0056583. Epub 2013 Feb 20. PMID 23437176